CLINICAL TRIAL: NCT03917953
Title: Transcutaneous Electrical Acupoint Stimulation for Treating Attention Deficit Hyperactivity Disorder: A Prospective, Randomized, Controlled Trial
Brief Title: Transcutaneous Electrical Acupoint Stimulation for the Treatment of ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xian Children's Hospital (Other Government); Shaanxi Hospital of Traditional Chinese Medicine (Other); Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2018-003
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Children with ADHD in the 2 groups were treated in separate treatment rooms and blinded on the intervention (i.e., true or sham TEAS). The TEAS operators could not be blinded to the treatment assignments. The data collectors, outcome assessors, and statisticians were blinded to group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive transcutaneous electrical acupoint stimulation therapy twice weekly for 4 weeks.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation
- Arm II (Sham Comparator): Patients receive sham transcutaneous electrical acupoint stimulation therapy twice weekly for 4 weeks.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Acupoint Stimulation — Patients in the experimental group will be treated for 20 min TEAS, twice a week, for a total of 4 weeks of treatment.The same intervention was performed in the sham group (electrode patches were attached at corresponding acupoints without electrical stimulation).
  Acupoint selection: baihui (GV 20), taichong (LR 3), taixi (KI 3).

SUMMARY:
RATIONALE: Transcutaneous electrical acupoint stimulation may improve attention deficit hyperactivity disorder (ADHD).

PURPOSE: This randomized-controlled trial study of treating attention deficit hyperactivity disorder of school-aged children with transcutaneous electrical acupoint stimulation to see how well it works compared to sham transcutaneous electrical acupoint stimulation.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

To determine whether true transcutaneous electrical acupoint stimulation(TEAS) administered twice weekly for 4 weeks (8 sessions) compared to sham TEAS causes a significant improvement in symptoms of ADHD according to the investigator-rated Clinical Global Impression-Improvement (CGI-I) scores at week 4.

Secondary

To evaluate the changes from baseline to week 4 of Clinical Global Impressions Scale-Severity of Illness (CGI-S)，Conners'Parent Rating Scales-Revised: Short Form (CPRS-R: S) score, Conners'Teacher Rating Scales-Revised: Short Form (CTRS-R: S) score, go/no-go task performances, and the concentration of oxygenated hemoglobin within the prefrontal cortex.

OUTLINE: This is a single-center study. Patients are randomized to two treatment arms.

Arm I: Patients receive TEAS twice weekly for 4 weeks . Arm II: Patients receive sham TEAS twice weekly for 4 weeks .

ELIGIBILITY:
Inclusion Criteria:

* Patients must be conform to ADHD clinical diagnostic criteria (DSM-V).
* Patients' ages are between 6~12 years old.
* An informed written consent from parents and participants

Exclusion Criteria:

* Patients have a history of illness that concomitant with other mental and neurological disorders.
* Patients's IQ score are lower than 75.
* Patients have had prior TEAS or other acupoints-associated treatment experiences.
* Left handedness.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
the investigator-rated Clinical Global Impression-Improvement (CGI-I) scores | 4 weeks
  The CGI-Improvement scale was used to evaluate the improvement, maintenance, or worsening of subjects' symptoms compared to baseline. The CGI-Improvement Scale includes seven options for scoring: 1 very much improved; 2 much improved; 3 minimally improved; 4 no change; 5 minimally worse; 6 much worse; and 7 very much worse. Clinical response at week 4 was defined as a rating of "much" or "very much improved" (1 or 2), which is considered a clinically meaningful response.

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement-Severity (CGI-S) score | 4 weeks
  The CGI-S includes seven options for scoring: 1 normal, not at all ill; 2 borderline mentally ill; 3 mildly ill; 4 moderately ill; 5 markedly ill; 6 severely ill; and 7 among the most extremely ill patients.
Conners' Parent Rating Scales-Revised: Short Form (CPRS-R: S) score | 4 weeks
  The CTRS-R:S is a teacher-rated 27-item 4-point Likert rating scale that contains items on ADHD and comorbid conditions (i.e., problems with conduct, emotion, anger control, and anxiety) in the home setting.
Conners' Teacher Rating Scales-Revised: Short Form (CTRS-R: S) score | 4 weeks
  The CTRS-R:S is a teacher-rated 28-item 4-point Likert rating scale that contains items on ADHD and comorbid conditions (i.e., problems with conduct, emotion, anger control, and anxiety) in the school setting.
go/no-go task performances | 4 weeks
  The accuracy (ACC) for go and no-go trials and reaction time (RT) of go trials were computed for each go/no-go block.
the concentration of oxygenated hemoglobin within the prefrontal cortex | 4 weeks
  fNIRS was used to monitor the brain response when the participants performed a go/no-go task before and after TEAS or sham TEAS treatment. The ETG-4000 (Hitachi Medical Corporation, Japan) multichannel fNIRS system to measure the relative concentration changes in oxygenated hemoglobin (HbO), with two wavelengths of nearinfrared light (695 and 830 nm). HbO signal is more sensitive to changes in cerebral blood flow than deoxygenated hemoglobin and total hemoglobin signals. Specifically, we used a 3 × 11 multichannel patch that consisted of 17 emitters and 16 detectors arranged alternately at an inter-probe distance of 3 cm forming 52 channels.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Dr., Principal Investigator — First Afflicated Hospital Xian Jiaotong University
Locations (1):
- Xian Children's Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Thapar A, Cooper M. Attention deficit hyperactivity disorder. Lancet. 2016 Mar 19;387(10024):1240-50. doi: 10.1016/S0140-6736(15)00238-X. Epub 2015 Sep 17. PMID 26386541
- [Background] Lee MS, Choi TY, Kim JI, Kim L, Ernst E. Acupuncture for treating attention deficit hyperactivity disorder: a systematic review and meta-analysis. Chin J Integr Med. 2011 Apr;17(4):257-60. doi: 10.1007/s11655-011-0701-7. Epub 2011 Apr 21. PMID 21509667
- [Background] Liu Z, Liu Y, Xu H, He L, Chen Y, Fu L, Li N, Lu Y, Su T, Sun J, Wang J, Yue Z, Zhang W, Zhao J, Zhou Z, Wu J, Zhou K, Ai Y, Zhou J, Pang R, Wang Y, Qin Z, Yan S, Li H, Luo L, Liu B. Effect of Electroacupuncture on Urinary Leakage Among Women With Stress Urinary Incontinence: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2493-2501. doi: 10.1001/jama.2017.7220. PMID 28655016
- [Background] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593
- [Derived] Zhuo L, Zhao X, Zhai Y, Zhao B, Tian L, Zhang Y, Wang X, Zhang T, Gan X, Yang C, Wang W, Gao W, Wang Q, Rohde LA, Zhang J, Li Y. Transcutaneous electrical acupoint stimulation for children with attention-deficit/hyperactivity disorder: a randomized clinical trial. Transl Psychiatry. 2022 Apr 21;12(1):165. doi: 10.1038/s41398-022-01914-0. PMID 35449191